CLINICAL TRIAL: NCT06399406
Title: Mindfulness Engaged Neurostimulation for Depression
Acronym: MEND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jyoti Mishra, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 809712
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Depression; Treatment Resistant Depression; Major Depressive Disorder; Depressive Disorder
Keywords: rTMS; mindfulness; depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Medi1-TBS (Experimental): This arm will receive a multimodal treatment with a digital mindfulness training focused on attention to breathing for up to 10 min session dose for up to 20 sessions combined with neuro-navigated iTBS type of rTMS (for 20 treatments over 4 weeks) targeting the left dorsolateral prefrontal cortex (DLPFC) brain region.
  Interventions: Combination Product: Medi-TBS
- Medi2-TBS (Experimental): This arm will receive a multimodal treatment with a digital mindfulness training focused on attention to breathing for up to 20 min session dose for up to 20 sessions combined with neuro-navigated iTBS type of rTMS (for 20 treatments over 4 weeks) targeting the left dorsolateral prefrontal cortex (DLPFC) brain region.
  Interventions: Combination Product: Medi-TBS
- Medi3-TBS (Active Comparator): This arm will receive a multimodal treatment with a digital mindfulness training focused on intermittent deep breathing for up to 10 min session dose for up to 20 sessions combined with neuro-navigated iTBS type of rTMS (for 20 treatments over 4 weeks) targeting the left dorsolateral prefrontal cortex (DLPFC) brain region.
  Interventions: Combination Product: Medi-TBS

INTERVENTIONS:
Combination Product: Medi-TBS — The multimodal intervention involves combining FDA-approved repetitive transcranial magnetic stimulation (rTMS) with digital mindfulness exercises.

SUMMARY:
Repetitive Transcranial Magnetic stimulation (rTMS) is an FDA-approved therapy for treatment resistant depression (TRD) that involves brief magnetic stimulation pulses on the dorsolateral prefrontal cortex (DLPFC) brain region. But studies of rTMS alone show remission rates of ~30%. Additionally, rTMS has not been shown to improve cognitive functioning that may be an independent factor predicting treatment success. This study will develop a novel multimodal treatment, which combines intermittent theta burst stimulation (iTBS) - a type of rTMS with digital mindfulness training to engage brain plasticity, enhance cognition and alleviate depression symptoms in individuals with TRD.

DETAILED DESCRIPTION:
This study aims to develop a novel multimodal treatment for treatment resistant depression (TRD), which combines intermittent theta burst stimulation (iTBS), a type of FDA-approved rTMS protocol, with digital mindfulness training. We propose that this multimodal treatment will suppress posterior Default Mode Network (pDMN) brain activity as measured with electroencephalography (primary outcome and neural target), as well as enhance cognition and alleviate depression symptoms in patients with TRD. The study will determine the optimal dose required for neural target engagement by the multimodal iTBS + digital mindfulness training relative to an active control training combined with iTBS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive episode (MDE, in accordance with the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5), in the context of unipolar major depressive disorder.
* At least one failed antidepressant medication trial at level 3 in the Antidepressant Treatment History Form: Short Form (ATHF-SF) classification.
* Montgomery-Åsberg Depression Rating Scale (MADRS) Score >19 (moderate - severe depression).
* No increase or initiation of new antidepressant therapy in the four weeks prior to screening.
* Demonstrated capacity to give informed consent.

Exclusion Criteria:

* Inability to provide informed consent.
* Medically unstable patients.
* Concomitant neurological disorder or a history of a seizure disorder.
* Exhibiting current suicidal behavior rating on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Patients who are pregnant or breastfeeding.
* Any psychotic disorder or current active psychotic symptoms.
* Patients who have intracranial implants, other medical device or condition deemed unsafe for TMS.
* Contraindication to MRI scanning.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in EEG source localized pDMN alpha activity | 4 weeks
  EEG alpha band (8-12 Hz) activity source-localized to the posterior Default Mode Network (pDMN) brain region extracted on distracted trials of the Breath Attention Assessment of Mindfulness task serves as the primary neural target.

SECONDARY OUTCOMES:
Change in Selective Attention | 4 weeks
  Processing speed of response to target stimuli on a standard continuous performance task that measures the ability to selectively attend and promptly respond to a goal-relevant target stimulus serves as the secondary cognitive target.
Change in Flanker Inhibition | 4 weeks
  Efficiency of inhibiting visuo-spatially flanking distractors to target stimuli in the Flanker task serves as the secondary cognitive target.
Change in Montgomery Åsberg Depression Rating Scale Scores (MADRS) | 8 weeks
  The MADRS will be used to evaluate % depressive symptom response defined as 50% change in the MADRS score from baseline as well as remission defined as MADRS score <7 at post-intervention. Scale range: 0-54, higher score is worse depression.

OTHER OUTCOMES:
Change in Working Memory | 4 weeks
  Span-weighted efficiency will be measured on a standard Delayed Match to Sample Task
Change in Mindful Attention Awareness Scale (MAAS) | 4 weeks
  The MAAS will be used to evaluate change in subjective state mindfulness. Scale range: 6-84, higher score is greater mindfulness
Change in Rumination Reflection Questionnaire (RRQ) | 4 weeks
  The RRQ will be used to evaluate change in subjective rumination. Scale range: 22-88, higher score is greater rumination
Change in Patient Health Questionnaire 9 item scale (PHQ9) | 8 weeks
  The PHQ9 scale will be used as an additional measure to evaluate change in depressive symptom response. Score range: 0-27, higehr score is greater depression
Change in Generalized Anxiety Disorder 7 item scale (GAD7) | 8 weeks
  The GAD7 scale will be used as a measure to evaluate change in anxiety symptom response.
  Score range: 0-21, higher score is greater anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mishra, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
In compliance with National Institute of Mental Health requirements for data sharing, collected data will be shared via the National Database for Clinical Trials related to Mental Illness (NDCT).
  Data submissions will include raw and processed data including basic demographic data, cognitive, behavioral, clinical data, and electroencephalography (EEG) data. All data will be structured as per a Data Dictionary that will be used for data harmonization purposes; data structure definitions will be taken from the existing NIMH Data Archive (NDA) Data Dictionary as recommended, however, if any data are not defined in the existing NDA Data Dictionary, then a new definition will be requested.
Time Frame: We will submit raw/descriptive data semi-annually (every January and July) and submit all other data at the time of publication of the initial report from the project.
Access Criteria: Access to study data will be available via the NDCT.

DOCUMENTS (1):
  • Informed Consent Form (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT06399406/ICF_000.pdf